CLINICAL TRIAL: NCT07384520
Title: Composition du Thrombus Dans Les Infarctus cérébraux : étude du Lien Avec Avec Des Biomarqueurs Plasmatiques, l'efficacité du Traitement, l'étiologie et le Pronostic.
Brief Title: Thrombus Composition in Cerebral Infarctions: Study of Its Association With Plasma Biomarkers, Treatment Efficacy, Etiology and Prognosis.
Acronym: COMPOCLOT
Status: Not yet recruiting | Type: Observational
Sponsor: François Delvoye (Other)
Responsible Party: Sponsor-Investigator, François Delvoye, Doctor, Centre Hospitalier Universitaire de Liege
Organization: Centre Hospitalier Universitaire de Liege (Other)
Other Study IDs: 2025-286
Record Dates: First submitted 2026-01-22; First posted 2026-02-03 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Ischemic Stroke; Cerebral Veinous Thrombosis
Keywords: Mechanical thrombectomy; Thrombus
MeSH Terms: conditions — Ischemic Stroke; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Thrombus, blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient treated with a thrombectomy

SUMMARY:
This study focuses on thrombi collected during mechanical thrombectomy procedures, as well as on plasma biomarkers analyzed concomitantly. The primary objective of the study is to investigate associations and correlations between, on the one hand, the composition of thrombi retrieved during thrombectomy and, on the other hand, plasma biomarkers, treatment response, etiology, and prognosis of ischemic stroke and cerebral venous thrombosis.

The secondary objectives of this study are to precisely characterize the biochemical composition of the thrombi (notably using techniques such as enzyme-linked immunosorbent assay [ELISA] following extraction of proteins contained within the thrombus), their histological structure (using standard histology with hematoxylin-eosin staining and immunohistochemistry), and their biological activity (in particular through in vitro assays assessing resistance to thrombolysis and the endothelial-adhesive or destructive properties of thrombi). Additional secondary objectives include testing new therapeutic methods for the lysis of thrombi collected by mechanical thrombectomy and establishing a link between thrombus transcriptomics and their confirmed etiology, particularly for thrombi initially described as having an embolic appearance and of undetermined etiology.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* Presenting with cerebral infarction secondary to an arterial occlusion responsible for an ischemic stroke, or with cerebral venous thrombosis (CVT) having undergone a mechanical thrombectomy (MT) procedure
* Managed with mechanical thrombectomy
* Provision of free, informed, and explicit consent by the patient or their legal representative/next of kin (emergency inclusion procedure)

Exclusion Criteria:

* Patients under legal protection measures (e.g., guardianship or curatorship)
* Patients for whom the thrombectomy specimen cannot be retrieved or is not suitable for analysis (estimated at approximately 50% of patients undergoing MT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Among patients treated at Liège University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2026-02-12 (Estimated); Primary Completion 2036-02-12 (Estimated); Study Completion 2036-05-30 (Estimated)

PRIMARY OUTCOMES:
Diminution or increase of the NIHSS (National Institutes of Health Stroke Scale) score. The scale goes from 0 to 42, the higher, the more severe. | In the 24 hours after the thrombectomy

IPD SHARING:
Plan to Share IPD: Undecided
Accessible upon request after publication

REFERENCES:
- [Background] Liebeskind DS, Sanossian N, Yong WH, Starkman S, Tsang MP, Moya AL, Zheng DD, Abolian AM, Kim D, Ali LK, Shah SH, Towfighi A, Ovbiagele B, Kidwell CS, Tateshima S, Jahan R, Duckwiler GR, Vinuela F, Salamon N, Villablanca JP, Vinters HV, Marder VJ, Saver JL. CT and MRI early vessel signs reflect clot composition in acute stroke. Stroke. 2011 May;42(5):1237-43. doi: 10.1161/STROKEAHA.110.605576. Epub 2011 Mar 10. PMID 21393591